CLINICAL TRIAL: NCT06546228
Title: Long Term Predictors of Acute Myocardial Infarction in Patients With Coronary Revascularization: a Machine Learning Analysis After a 7 Years Follow-up
Brief Title: Long Term Predictors of Acute Myocardial Infarction in Patients With Coronary Revascularization
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Other Study IDs: 01-21
Record Dates: First submitted 2024-07-12; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Acute Myocardial Infarction; Revascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention. Only observational. — Only collection of data or parameters already required by the medical examination programmed.

SUMMARY:
Worldwide, Ischemic heart disease is the single most common fatal disease. One of the most common causes of acute myocardial infarction is represented by obesity. Numerous cardio metabolic variables play a key role in incidence of adverse cardiovascular outcomes. The purpose of this research was to investigate the factors allowing to acute coronary syndrome, related to the metabolic status, to help guide each patient toward early preventing behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Patients met the criteria for Acute Coronary Syndrome (ACS) as defined by the Joint European Society of Cardiology/American College of Cardiology Committee.
* Patients underwent immediate coronary revascularization (primary PCI) for ST-Elevation Myocardial Infarction (STEMI).
* Patients underwent coronary revascularization (early PCI) within 24 hours for Non-ST-Elevation Myocardial Infarction (NSTEMI).
* Patients underwent diagnostic coronary angiography following coronary artery bypass graft surgery (CABG).

Exclusion Criteria:

* Known coronary artery disease or previous ACS.
* PCI following CABG.
* Cardiogenic shock.
* Atrial fibrillation.
* Peripheral artery disease.
* Severe cardiac valve disease.
* Prosthetic aorta.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized for acute coronary syndrome (ACS)
Sampling Method: Non-Probability Sample
Enrollment: 652 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Acute Myocardial Infarction (AMI) | 7 years
  Occurrence of AMI. Unit of measure: Medical records, electrocardiogram (ECG), cardiac biomarkers

SECONDARY OUTCOMES:
Change in Left Ventricular Ejection Fraction (LVEF) | 7 years
  LVEF before and after revascularization Measurement Tool: Echocardiogram Unit of Measure: Percentage (%) change in LVEF
Incidence of Cardiovascular Death | 7 years
  Occurrence of cardiovascular death Measurement Tool: Medical records Unit of Measure: Number of cardiovascular deaths per patient-year

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria G. Martino, Messina, Italy

IPD SHARING:
Plan to Share IPD: No
Anonymous data